CLINICAL TRIAL: NCT06606054
Title: WSO - The Brain and hEart globAl iniTiative (BEAT) Stroke
Brief Title: WSO BEAT STROKE Initiative
Acronym: BEAT STROKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: W.L.Gore & Associates (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14852
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stroke; PFO - Patent Foramen Ovale; Atrial Fibrillation (AF)
Keywords: cardiac monitoring; stroke; atrial fibrillation; pfo closure
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No intervention (Placebo Comparator): This group will not receive any of the educational and/or implementation Neurocardiology until the data collection is completed.
  Interventions: Other: No educational or implementation tool will be provided
- Intervention arm (Active Comparator): Sites randomized in this arm will receive the educational and implementation Neurocardiology tool with the aim of improving adherence to best practice recommendations for secondary stroke prevention of cardioembolic strokes, as defined by the WSO Systematic Review and Synthesis of Global Stroke Guidelines or more recent high-quality evidence published after the last stroke guidelines.
  Interventions: Other: Educational and implementation Neurocardiology tool

INTERVENTIONS:
Other: Educational and implementation Neurocardiology tool — Sites in this arm will be provided with an educational and implementation Neurocardiology tool aiming to improve adherence to best practice recommendations for secondary stroke prevention of cardioembolic strokes, as defined by the WSO Systematic Review and Synthesis of Global Stroke Guidelines or more recent high-quality evidence published after the last stroke guidelines1.
  Arms: Intervention arm
Other: No educational or implementation tool will be provided — Participants will be followed for up to 12 months. No educational or interventional tool will be provided to sites in this arm until the follow-up period has ended.
  Arms: No intervention

SUMMARY:
The WSO Brain and hEart globAl iniTiative - STROKE (BEAT-STROKE) is a cluster randomized controlled trial, testing whether an educational and implementation Neurocardiology tool can improve adherence to best practice recommendations for secondary stroke prevention of cardioembolic strokes, as defined by the WSO Systematic Review and Synthesis of Global Stroke Guidelines or more recent high-quality evidence published after the last stroke guidelines1

DETAILED DESCRIPTION:
The World Stroke Organization (WSO) Brain and Heart Task Force developed The Brain & hEart globAl iniTiative (BEAT), a pilot feasibility program aimed at establishing clinical collaborations between cardiologists and stroke physicians.1 The WSO BEAT pilot project focused on atrial fibrillation (AF) and patent foramen ovale (PFO) detection and management, highly prevalent cardioembolic causes of ischemic stroke and transient ischemic attack (TIA).

The pilot feasibility WSO BEAT program comprised 10 sites from 8 countries, including Brazil, China, Egypt, Germany, Japan, Mexico, Romania, and the USA. Of the 10 sites, two belonged exclusively to the public sector and one was public and private. The primary objective of the pilot WSO BEAT program was to assess its feasibility by achieving a composite feasibility outcome including: (1) developing site-specific clinical pathways for the diagnosis and management of AF, PFO, and the stroke heart syndrome; (2) establishing regular Neurocardiology rounds (e.g., monthly, bimonthly, etc.); and (3) incorporating a cardiologist to the stroke team.

Overall, the WSO BEAT program successfully achieved the pre-specified goals at most sites. Regarding the three primary program objectives, 9/10 (90%) of the sites were able to design or update the proposed clinical care pathways, establish Neurocardiology rounds, and designate a dedicated cardiologist for the stroke team, respectively.

To date it is unknown whether the implementation of Neurocardiology educational tools and collaborations between cardiologists and neurologists can improve adherence to best practice recommendations focused on the management of cardioembolic strokes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke or TIA of any etiology.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference between the baseline and 6-month mean WSO BEAT Neurocardiology Score | 6-months
  Difference between the baseline and 6-month mean WSO BEAT Neurocardiology Score. The score for each patient will be calculated by adding the total points and dividing this number by the total ideal points for that patient, given that not all patients will qualify for the (embolic stroke of undetermined source (ESUS), PFO or AF points).

SECONDARY OUTCOMES:
Difference between the baseline and 6-month mean WSO BEAT Neurocardiology Score for each of the 5 pre-specified cathegories. | 6-months
  Difference between the baseline and 6-month mean WSO BEAT Neurocardiology Score for each of the 5 pre-specified categories: basic assessment, stroke-heart syndrome, ESUS workup, PFO in young patients, and AF management.
Long-term achievement of the primary outcome at 12 months. | 12-months
  Difference between the baseline and 12-month mean WSO BEAT Neurocardiology Score. The score for each patient will be calculated by adding the total points and dividing this number by the total ideal points for that patient, given that not all patients will qualify for the (embolic stroke of undetermined source (ESUS), PFO or AF points).

OTHER OUTCOMES:
Exploratory endpoint. Major adverse cardiovascular events (MACE) at 12 months | 12-months
  Major adverse cardiovascular events (MACE) at 12 months defined as the composite of the following events:
  * Recurrent ischemic stroke.
  * Acute coronary event.
  * Admission or Emergency Department visit for decompensated heart failure (HF), AF, or valvular heart disease.
  * New diagnosis of coronary artery disease.
  * Cardiovascular death.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart & Brain Lab, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request and after the Approval of Western University Ethics Review Board